CLINICAL TRIAL: NCT05371054
Title: Phase 1/2 Study of VIP152, Venetoclax, and Prednisone (VVIP) in Relapsed/Refractory Lymphoid Malignancies
Brief Title: Study of VIP152, Venetoclax, and Prednisone (VVIP) in Relapsed/Refractory Lymphoid Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Melani, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000633; 000633-C
Record Dates: First submitted 2022-05-11; First posted 2022-05-12 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma; Non-Hodgkin Lymphoma; NHL; Hematologic Malignancies; Lymphoid Malignancies
Keywords: Dose Finding; Small Molecule
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Hematologic Neoplasms | interventions — venetoclax; Prednisone; Positron-Emission Tomography; Electrocardiography; Echocardiography; Magnetic Resonance Imaging; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1/Phase 1: Arm 1 Dose Escalation (Experimental): Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Interventions: Device: Vysis LSI MYC Break Apart Rearrangement Probe Kit; Drug: Venetoclax; Drug: VIP152; Drug: Prednisone; Diagnostic Test: PET; Diagnostic Test: EKG; Diagnostic Test: ECHO; Diagnostic Test: CT neck chest, abdomen, and pelvis; Diagnostic Test: MRI; Procedure: Bone marrow aspiration/Biopsy
- Cohort 2/Phase 2: Arm 2 Dose Expansion (Experimental): Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at the recommended phase II dose (RP2D) with prednisone at fixed doses.
  Interventions: Device: Vysis LSI MYC Break Apart Rearrangement Probe Kit; Drug: Venetoclax; Drug: VIP152; Drug: Prednisone; Diagnostic Test: PET; Diagnostic Test: EKG; Diagnostic Test: ECHO; Diagnostic Test: CT neck chest, abdomen, and pelvis; Diagnostic Test: MRI; Procedure: Bone marrow aspiration/Biopsy

INTERVENTIONS:
Device: Vysis LSI MYC Break Apart Rearrangement Probe Kit — MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
Drug: Venetoclax — Dose Escalation: Administered orally, days 1-10, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity.
  Dose Expansion: Administered orally, days 1-10, at the recommended phase 2 dose (RP2D); every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Other Names: Venclexta; Venclyxto
Drug: VIP152 — Dose Escalation: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity.
  Dose Expansion: Administered intravenously, days 2 and 9, at the recommended phase 2 dose (RP2D); every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity.
  Other Names: Enitociclib
Drug: Prednisone — Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Other Names: Rayos; Deltasone; Prednisone Intensol
Diagnostic Test: PET — Screening, pre-cycle 7, pre-cycle 13, and at end-of-treatment (post-cycle 24).
  Other Names: Positron emission imaging
Diagnostic Test: EKG — Screening
  Other Names: Electrocardiogram
Diagnostic Test: ECHO — Screening
  Other Names: Echocardiogram
Diagnostic Test: CT neck chest, abdomen, and pelvis — Screening, pre-cycle 2, pre-cycle 3, pre-cycle 5, pre-cycle 7, pre-cycle 9, pre-cycle 11, pre-cycle 13, pre-cycle 15, pre-cycle 17, pre-cycle 19, pre-cycle 21, pre-cycle 23, and at end-of-treatment (post cycle 24).
  Other Names: Computed tomography neck chest, abdomen, and pelvis
Diagnostic Test: MRI — As indicated. Screening, pre-cycle 2, pre-cycle 3, pre-cycle 5, pre-cycle 7, pre-cycle 9, pre-cycle 11, pre-cycle 13, pre-cycle 15, pre-cycle 17, pre-cycle 19, pre-cycle 21, pre-cycle 23, and at end-of-treatment (post cycle 24).
  Other Names: Magnetic resonance imaging
Procedure: Bone marrow aspiration/Biopsy — Baseline, post-cycle 6, post-cycle 12, and at end-of-treatment (post-cycle 24).
  Other Names: BM aspiration/Bx

SUMMARY:
Background:

Non-Hodgkin lymphomas are blood cancers that can be difficult to treat. They can also return after treatment. Examples include diffuse large B-cell lymphoma (DLBCL) and peripheral T-cell lymphoma (PTCL). More effective treatments are needed for these diseases.

Objective:

To test the safety of a study drug (Enitociclib (VIP152) in combination with other drugs used to treat people with aggressive blood cancers.

Eligibility:

People aged 18 years or older diagnosed with DLBCL, PTCL, or related blood cancers. The cancers must have either not responded to treatment or returned after treatment.

Design:

Participants will undergo screening. They will have a physical exam with scans and blood and urine tests. They will have imaging scans and tests of their heart function. They may also provide a bone marrow aspiration or biopsy.

Participants may provide a saliva sample for deoxyribonucleic acid (DNA) testing.

Participants will receive study treatment in cycles. Each cycle is 21 days.

Participants will take two drugs by mouth at home once a day on days 1-10 of each cycle.

On days 2 and 9 they will come to the clinic to receive VIP152. This drug will be administered through a small plastic tube with a needle placed in a vein.

On day 11, participants will receive a fourth medication as an injection under the skin. They will rest and recover on days 12-21.

Screening tests will be repeated periodically throughout the study period.

Treatment will continue for up to 24 cycles.

Participants will have follow-up visits for up to 5 years.

DETAILED DESCRIPTION:
Background:

* High unmet medical need for relapsed/refractory non-Hodgkin lymphoma (NHL) after exhausting chemotherapy and/or chemo-immunotherapy regimens
* Targeted therapies aimed at disrupting cell death pathway in hematologic malignancies are emerging and showing significant activity in both the relapsed and first-line settings
* Enitociclib (VIP152) is a selective inhibitor of positive transcription elongation factor (PTEFb)/Cyclin-dependent kinase 9 (CDK9) and is expected to show efficacy in tumor indications that overexpress MYC and myeloid Cell Leukemia-1 (MCL-1). VIP152 monotherapy has demonstrated a mild toxicity profile and preliminary efficacy in Phase 1 studies in advanced cancer
* The combination of VIP152 with venetoclax and prednisone (VVIP) targets major cell-death pathways in lymphoid malignancies (B-cell lymphoma 2 (BCL-2 and myeloid cell leukemia 1 (MCL-1) and may overcome chemo-resistance and/or single drug resistance to venetoclax.

Objectives:

* Phase 1: To determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), and the safety and toxicity profile of the combination of VIP152 with venetoclax and prednisone (VVIP) in relapsed/refractory lymphoid malignancies
* Phase 2: To determine the complete response (CR) rate of the combination of VIP152 with venetoclax and prednisone (VVIP) in R/R lymphoid malignancies

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have a histologically or cytologically confirmed lymphoid malignancy as listed below, confirmed by the Laboratory of Pathology, National Cancer Institute (NCI), as follows:

  * Refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/High-grade B-cell lymphoma (HGBCL) (MYC aberration must be confirmed by NCI Laboratory of Pathology to enroll)
  * R/R non-germinal center B-cell (non-GCB) DLBCL without MYC-rearrangement (Cell of origin (COO) and non-MYC aberration must be confirmed by NCI Laboratory of Pathology to enroll. COO determination at enrollment will utilize immunohistochemistry and Han's algorithm)
  * R/R Peripheral T-cell lymphoma (PTCL-not otherwise specified (NOS), PTCL-T follicular helper (TFH), follicular T-cell lymphoma (TCL), angioimmunoblastic T-cell lymphoma (AITL), adult T-cell leukemia/lymphoma (ATLL), anaplastic lymphoma kinase (ALK)+ anaplastic large-cell lymphoma (ALCL) and ALK- ALCL per 2016 World Health Organization (WHO) classification)
* Relapsed and/or refractory disease, as defined below:

  * Aggressive B-cell lymphoma: relapsed after and/or refractory to at least 2 prior systemic therapies, 1 or more which includes an anthracycline and anti-cluster of differentiation 20 (CD20) targeting agent
  * PTCL: relapsed after and/or refractory to at least 2 prior systemic therapies, 1 or more which includes an anthracycline (and a brentuximab vedotin-containing regimen for participants with ALK+ or ALK- ALCL)
* Must have evaluable disease by clinical exam (i.e., palpable lymphadenopathy, measurable skin lesions, etc.), laboratory assessment (i.e., disease involvement of bone marrow or peripheral blood by morphology, cytology or flow cytometry), and/or imaging (measurable lymph nodes, masses, or bony lesions on computed tomography (CT) or magnetic resonance imaging (MRI) and/or evaluable FD-Gavid lesions on positron emission tomography (PET).

NOTE: Lesions that have been irradiated cannot be included in the tumor assessment unless unequivocal tumor progression has been documented in these lesions after radiation therapy.

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2
* Adequate organ and marrow function as defined below unless dysfunction is secondary to disease:

  * Absolute neutrophil count* >=1,000/mcL
  * Hemoglobin* >=8 g/dL
  * Platelets >=75,000/mcL
  * International normalized ratio (INR) <=1.5 X institutional upper limit of normal (ULN) for participants not receiving therapeutic anticoagulation
  * Partial thromboplastin time (PTT)/activated partial thromboplastin time (aPTT) <= 1.5 X institutional ULN normal except if the aPTT is elevated because of a positive Lupus Anticoagulant
  * Total bilirubin** <=1.5 X institutional ULN (or <=3 X institutional ULN for participants with documented Gilbert's syndrome)
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)(SGOT)/Alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT)*** <= 2.5 X institutional ULN
  * Serum creatinine <= 2.0 mg/dL

OR

--Creatinine clearance**** >= 40 mL/min/1.73 m^2 for participants with creatinine levels above 2 mg/dL

Creatinine clearance (Cr Cl) will be calculated with the use of the 24-hour creatinine clearance or modified

Cockcroft-Gault equation (eCCR; with the use of ideal body mass [IBM] instead of mass): (140 - Age) x IBM (kg) x [0.85 if female] / 72 x serum creatinine (mg/dL)

*Red blood cell (RBC) transfusions and use of granulocyte colony-stimulating factor (G-CSF) will be allowed in order to meet eligibility parameters.

* Total bilirubin must be <= 3 X institutional ULN for eligibility even if secondary to disease.

  * AST(SGOT)/ALT(SGPT) must be <= 5 X institutional ULN for eligibility even if secondary to disease.

    * Creatinine clearance must be >= 30 mL/min for eligibility even if secondary to disease.

      * Negative serum or urine pregnancy test must be obtained within 7 days before the first dose of study drug in individuals of childbearing potential. Postmenopausal individuals, as defined below, are allowed to enroll without a pregnancy test:

        --Age >50 years with amenorrhea for at least 12 months or

        --Age <=50 years with 6 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) level within postmenopausal range (>40 mIU/mL) OR
        * Permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, uterine ablation)
      * Individuals of reproductive potential must agree to use highly effective contraception when sexually active. This applies for the period between signing of the informed consent and 90 days after the last administration of study drug.

Highly effective contraception includes:

* Established use of oral, injected or implanted hormonal methods of contraception
* Placement of certain intrauterine devices (IUD) or intrauterine systems (IUS)
* Hysterectomy, oophorectomy, salpingectomy or vasectomy of the partner (provided that partner is the sole sexual partner of the individual of childbearing potential trial participant and that the vasectomized partner has received medical assessment of the surgical success)

In addition, participants must agree to use condoms.

* Participants that are positive for hepatitis B core antibody (HBcAb), hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb) must have a negative hepatitis B and/or C viral load by polymerase chain reaction (PCR), and agree to additional monitoring.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Nursing participants must be willing to discontinue nursing from study treatment initiation through 90 days after the last administration of study drug.

EXCLUSION CRITERIA:

-The following restrictions apply to current or prior anti-cancer treatment, prior to the first dose of study drug:

* Participants who are actively receiving any other anti-cancer investigational agents.
* Any chemotherapy, targeted therapy, or anti-cancer antibodies within 2 weeks prior to the first dose of study drug
* Radio- or toxin-immunoconjugates within 10 weeks prior to the first dose of study drug
* Prior allogeneic stem cell (or other organ) transplant within 6 months or any evidence of active graft-versus-host disease or requirement for immunosuppressants within 28 days prior to first dose of study drug
* Not recovered (i.e., <= Grade 1 or baseline) from adverse events due to previously administered anti-cancer treatment, surgery, or procedure.

NOTE: Exceptions to this include events not considered to place the participant at unacceptable risk of participation in the opinion of the principal investigator (PI) (e.g., alopecia).

-Participants requiring the following agents within 14 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of venetoclax and VIP152 are excluded:

* Strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors
* Strong CYP3A inducers
* Moderate CYP3A inhibitors (dose-escalation cohort only)
* Moderate CYP3A inducers (dose-escalation cohort only)

NOTE: Moderate CYP3A inhibitors and inducers should be used with caution for participants in the dose-expansion cohorts and an alternative medication used, whenever possible.

* Known allergy to both xanthine oxidase inhibitors and rasburicase; or known hypersensitivity to any of the study drugs
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 2 weeks prior to first dose of study drug
* HIV-positive participants
* Active cytomegalovirus (CMV) infection as determined by a positive CMV polymerase chain reaction (PCR)
* Active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection based on PCR assay; prior SARs-CoV-2 infection allowed if completely recovered from infection and negative PCR testing
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis; as well as active infection with hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) except as noted above in inclusion criteria

  * Participants with occult or prior HBV infection (defined as positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (HBcAb)) may be included if HBV deoxyribonucleic acid (DNA) is undetectable (i.e., none detected in copies/mL or IU/mL). These individuals must be willing to undergo HBV DNA testing during treatment and in surveillance for at least 12 months after completion of study therapy.
  * Participants who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
* Malabsorption syndrome or other condition that precludes enteral route of administration
* History of other active malignancy requiring therapy that could affect compliance with the protocol or interpretation of results
* Symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Left ventricular ejection fraction (LVEF) < 45%
* Clinically relevant findings on electrocardiogram (ECG) such as a second- or third-degree AV block or prolongation of the heart-rate corrected QT interval (Qtc) (Fridericia) over 470 msec (participants with atrioventricular (AV) block and pacemaker in place for >1 year and checked by a cardiologist within <6 months before the first dose of study drug, will not be excluded).
* Uncontrolled intercurrent illness (including psychiatric) or social situations that may limit interpretation of results or that could increase risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Melani, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. Genomic data will be available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data will be made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Frigault MM, Mithal A, Wong H, Stelte-Ludwig B, Mandava V, Huang X, Birkett J, Johnson AJ, Izumi R, Hamdy A. Enitociclib, a Selective CDK9 Inhibitor, Induces Complete Regression of MYC+ Lymphoma by Downregulation of RNA Polymerase II Mediated Transcription. Cancer Res Commun. 2023 Nov 9;3(11):2268-2279. doi: 10.1158/2767-9764.CRC-23-0219. PMID 37882668
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000633-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP)-VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL), R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg; Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL, R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 4 Enitociclib (VIP152) 30mg & Venetoclax 800mg: No participants were enrolled in cohort 1/phase 1:Arm 1 dose escalation dose level 4. VIP152, Venetoclax, & prednisone-Enitociclib(VIP152) & venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose & recommended phase II dose of VIP152 & venetoclax. Vysis LSI MYC Break Apart Rearrangement Probe Kit:MYC rearrangement fluorescence in situ hybridization testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research, National Cancer Institute. This kit is not Food and Drug Administration approved. It is being used as a treatment determining in-vitro diagnostic device in this study. Venetoclax:Administered orally, days 1-10, per specified dose level;every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity. VIP152:Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity. Prednisone:Administered orally, days 1-10, at a dose of 100mg;every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity. Cohort 1 Dose Escalation:participants with either refractory/relapsed (R/R)MYC-rearranged diffuse large B-cell lymphoma/high-grade B-cell lymphoma, R/R non-germinal center B-Cell diffuse large B-cell lymphoma(no MYC rearrangement) &/or R/R peripheral T-cell lymphoma.
- Cohort 2/Phase 2: Arm 2 Dose Expansion with Enitociclib (VIP152) & Venetoclax: No participants were enrolled in cohort 2/phase 2: Arm 2 dose expansion.
  Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at the recommended phase II dose (RP2D) with prednisone at fixed doses.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, at the recommended phase 2 dose (RP2D); every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, at the recommended phase 2 dose (RP2D); every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Participants with refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL) for Phase 2 dose expansion.
Period: Overall Study
Arm/Group | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 4 Enitociclib (VIP152) 30mg & Venetoclax 800mg | Cohort 2/Phase 2: Arm 2 Dose Expansion with Enitociclib (VIP152) & Venetoclax
Started | 3 | 3 | 2 | 0 | 0
Completed | 3 | 3 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 24 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL), R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
- Total: Total of all reporting groups
Arm/Group | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg | Total
Number analyzed (Participants) | 3 | 3 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 5
  >=65 years | 1 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.67 (12.42) | 68.33 (12.22) | 43.5 (6.36) | 60 (14.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 2 | 3 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 1 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Complete Response (CR) Rate
Description: CR rate is defined as the percentage of participants who meet criteria for complete response (CR) as measured by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL). Complete response is defined as target nodes/nodal masses that regress to <1.5 cm in longest transverse diameter of a lesion (LDi).
Time Frame: 24 cycles (i.e., 72 weeks)
Population: This outcome measure was not done because no participants were enrolled in the phase 2 cohort.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 2/Phase 2: Arm 2 Dose Expansion with Enitociclib (VIP152) & Venetoclax: No participants were enrolled in cohort 2/phase 2: Arm 2 dose expansion. Enitociclib (VIP152), Venetoclax, and prednisone (VVIP) - VIP152 and venetoclax at the recommended phase II dose (RP2D) with prednisone at fixed doses.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose levelat the RP2D; every 21 days for up to 12 24 cycles, or until disease progression or unacceptable toxicity VIP152: Administered intravenously, days 2 and 9, per specified dose levelat the RP2D; every 21 days for up to 12 24 cycles, or until disease progression or unacceptable toxicity Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 24 cycles, or until disease progression or unacceptable toxicity Participants with refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL) for Phase 2 dose expansion.
Arm/Group | Cohort 2/Phase 2: Arm 2 Dose Expansion with Enitociclib (VIP152) & Venetoclax
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 1: Number of Solicited and/or Non-solicited Non-serious Adverse Events (AE's) With Grade
Description: Number of non-serious adverse events (AE's) with grade was assessed by the CTCAEv5.0. A non-serious adverse event is any untoward medical occurrence that does not meet seriousness criteria. Grade 1 is mild. Grade 2 is moderate. Grade 3 is serious. Grade 4 if life-threatening.
Time Frame: Up to 18 weeks.
Measure: Number; unit: adverse events
Groups:
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL), R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg: Venitociclib (VIP152), venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL, R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL, R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
Arm/Group | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
adverse events
  Grade 1 Alanine aminotransferase increased | 0 | 0 | 1
  Grade 1 Alkaline phosphatase increased | 2 | 4 | 1
  Grade 1 Anemia | 9 | 7 | 3
  Grade 1 Aspartate aminotransferase increased | 0 | 0 | 1
  Grade 1 Blood bilirubin increased | 0 | 0 | 1
  Grade 1 Bone pain | 0 | 1 | 0
  Grade 1 Constipation | 0 | 1 | 0
  Grade 1 Creatinine increased | 0 | 0 | 2
  Grade 1 Cytomegalovirus infection reactivation | 1 | 4 | 0
  Grade 1 Diarrhea | 1 | 2 | 0
  Grade 1 Edema limbs | 1 | 0 | 0
  Grade 1 Fatigue | 2 | 0 | 0
  Grade 1 Flatulence | 1 | 0 | 0
  Grade 1 Headache | 0 | 1 | 0
  Grade 1 Hypokalemia | 0 | 1 | 0
  Grade 1 Hypomagnesemia | 3 | 4 | 0
  Grade 1 Insomnia | 1 | 0 | 0
  Grade 1 Nausea | 1 | 0 | 0
  Grade 1 Neutrophil count decreased | 0 | 4 | 1
  Grade 1 Pain in extremity | 1 | 0 | 0
  Grade 1 Platelet count decreased | 7 | 9 | 4
  Grade 1 Rash maculopapular | 1 | 1 | 0
  Grade 1 Skin and subcutaneous tissue disorders - tinea corporis | 0 | 1 | 0
  Grade 2 Anemia | 6 | 6 | 1
  Grade 2 Back pain | 0 | 1 | 0
  Grade 2 Creatinine increased | 0 | 0 | 2
  Grade 2 Hyperphosphatemia | 0 | 0 | 1
  Grade 2 Hypokalemia | 5 | 4 | 1
  Grade 2 Neutrophil count decreased | 3 | 4 | 0
  Grade 2 Pain in extremity | 1 | 0 | 0
  Grade 2 Platelet count decreased | 0 | 2 | 1
  Grade 2 Skin infection | 1 | 0 | 0
  Grade 3 Hypokalemia | 1 | 0 | 0
  Grade 3 Neutrophil count decreased | 2 | 1 | 0
  Grade 3 Platelet count decreased | 0 | 1 | 0
  Grade 4 Neutrophil count decreased | 0 | 4 | 1

3. Primary Outcome: Phase 1: Number of Solicited and/or Unsolicited Serious Adverse Events (SAE's) With Grade
Description: Number of serious adverse events (SAE's) with grade was assessed by the CTCAEv5.0. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is fatal.
Time Frame: Up to 18 weeks.
Measure: Number; unit: Adverse events
Groups:
- Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg; Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL, R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
Arm/Group | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg & Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Adverse events
  Grade 2 Lymph node pain | 0 | 1 | 0
  Grade 3 Alanine aminotransferase increased | 0 | 0 | 1
  Grade 3 Aspartate aminotransferase increased | 0 | 0 | 1

4. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D)
Description: The MTD/RP2D is the dose level at which no more than 1 of up to 6 participants experience dose limiting toxicity (DLT) during the DLT evaluation window(s), or the dose below that at which at least 2 (of ≤6) participants have DLT. A DLT (dose-limiting toxicity) is defined as a grade 3 or higher adverse event (AE) that occurs in the dose-escalation cohort within the first 22 days after initiation of VVIP (i.e., Cycle 1, Day 1 to Cycle 2, Day 1 pre-dose) and is considered related to study drug (i.e., VIP152, venetoclax, and/or prednisone) or a treatment delay of cycle 2 of > 7 days for hematologic or nonhematologic toxicities.
Time Frame: First 22 days (i.e., cycle 1, day 1 to cycle 2, day 1 pre-dose)
Measure: Number; unit: mg
Groups:
- All Participants: All participants who received at least one dose of any study agent and completed the dose-limiting toxicity (DLT) evaluation window.
Arm/Group | All Participants
Number analyzed (Participants) | 8
mg | NA — MTD/RP2D was not found because the study was prematurely closed.

5. Primary Outcome: Phase 1: Number of Participants With Grade 4 Neutropenia Dose-Limiting Toxicity (DLT)
Description: A DLT (dose-limiting toxicity) is defined as a grade 3 or higher adverse event (AE) that occurs in the dose-escalation cohort within the first 22 days after initiation of VVIP (i.e., Cycle 1, Day 1 to Cycle 2, Day 1 pre-dose) and is considered related to study drug (i.e., VIP152, venetoclax, and/or prednisone) or a treatment delay of cycle 2 of > 7 days for hematologic or nonhematologic toxicities.
Time Frame: First 22 days (i.e., cycle 1, day 1 to cycle 2, day 1 pre-dose)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL), R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
- Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg: Enitociclib (VIP152), Venetoclax and prednisone (VVIP) - VIP152 and venetoclax at escalating doses with prednisone at fixed doses to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of VIP152 and venetoclax.
  Vysis LSI MYC Break Apart Rearrangement Probe Kit: MYC rearrangement fluorescence in situ hybridization (FISH) testing is performed using the Vysis LSI MYC Break Apart Rearrangement Probe (Abbott Molecular, Inc.) in the Chromosome Pathology Section, Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). This kit is not Food and Drug Administration (FDA) approved. It is being used as a treatment determining in-vitro diagnostic device in this study.
  Venetoclax: Administered orally, days 1-10, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  VIP152: Administered intravenously, days 2 and 9, per specified dose level; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Prednisone: Administered orally, days 1-10, at a dose of 100 mg; every 21 days for up to 12 cycles, or until disease progression or unacceptable toxicity
  Cohort 1 Dose Escalation: participants with either refractory/relapsed (R/R) MYC-rearranged diffuse large B-cell lymphoma (DLBCL)/high-grade B-cell lymphoma (HGBCL, R/R non-germinal center B-Cell (GCB) DLBCL (no MYC rearrangement) and/or R/R peripheral T-cell lymphoma (PTCL)
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Participants | 0 | 0 | 1

6. Secondary Outcome: Phase 1: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from the date of study enrollment until the date of disease relapse, disease progression, death, or last follow-up, whichever occurs first, using the Kaplan-Meier method. Response was assessed by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL). Disease progression is defined as an increase of ≥ 50% from the product of the perpendicular diameter (PPD) nadir and an increase in longest transverse diameter of a lesion (LDi) or shortest axis perpendicular diameter (SDi) from nadir of >0.5 cm for lesions <2 cm or >1.0 cm for lesions >2 cm.
Time Frame: Assessed from date of study enrollment until time of disease relapse, disease progression, death, or last follow-up, whichever comes first, up to 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Months | 1.48 [0.49 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | 4.14 [2.99 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | 4.11 [2.14 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable.

7. Secondary Outcome: Phase 1: Time to Response (TTR)
Description: TTR is defined as the time from the start of the treatment until time of first objective response using the Kaplan-Meier method. Median, assessed during therapy and after completion of therapy from initiation of therapy to first response every (q)3, 4, 6 and 12 months for post-treatment years 1, 2, 3, and 4-5, respectively, for up to 5 years after the last participant has enrolled on study. Response was measured by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL). Complete response is target nodes/nodal masses that regress to <1.5 cm in longest transverse diameter of a lesion. Partial response is ≥ 50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of up to 6 target measurable nodes and extranodal sites. Disease progression is an increase by ≥ 50% from progressive disease progression (PPD) nadir and an increase in longest transverse diameter of a lesion (LDi) or shortest axis perpendicular diameter (SDi) from nadir.
Time Frame: Time from the date of study enrollment during therapy, after completion of therapy from initiation of therapy to first response, up to 5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Months | 3.45 [NA to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | 0.69 [0.66 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | NA [NA to NA] — Median and 95% confidence interval is not estimable because not evaluable since no responses.

8. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR is defined as the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented using the Kaplan-Meier method. Response was measured by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL). Complete response is target nodes/nodal masses that regress to <1.5 cm in longest transverse diameter of a lesion (LDi). Partial response is ≥ 50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of up to 6 target measurable nodes and extranodal sites. Disease progression is an increase by ≥ 50% from progressive disease progression (PPD) nadir and an increase in longest transverse diameter of a lesion (LDi) or shortest axis perpendicular diameter (SDi) from nadir of >0.5 cm for lesions <2 cm or >1.0 cm for lesions >2 cm.
Time Frame: Time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Months
  Complete Response | NA [NA to NA] — Median and 95% confidence interval cannot be calculated since none of these participants achieved a response. | NA [NA to NA] — Median and 95% confidence interval cannot be calculated since none of these participants achieved a response. | NA [NA to NA] — Median and 95% confidence interval cannot be calculated since neither of these participants achieved a response.
  Partial Response | 4.37 [NA to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | 3.45 [2.33 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | NA [NA to NA] — Median and 95% confidence interval cannot be calculated since neither of these participants achieved a response.

9. Secondary Outcome: Phase 1: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants who meet criteria for complete response (CR) or partial response (PR) as measured by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL). Complete response is target nodes/nodal masses that regress to <1.5 cm in longest transverse diameter of a lesion (LDi). Partial response is ≥ 50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of up to 6 target measurable nodes and extranodal sites.
Time Frame: 24 cycles (i.e., 72 weeks)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Proportion of participants
  Complete Response | 0 [0 to 0.708] | 0 [0 to 0.708] | 0 [0 to 0.842]
  Partial Response | 0.3333 [0.0084 to 0.9057] | 1.000 [0.292 to 1.000] | 0 [0 to 0.842]

10. Secondary Outcome: Phase 1: Overall Survival (OS)
Description: OS is defined as the time from the date of study enrollment until death from any cause, or last follow-up, whichever occurs first, assessed using the Kaplan-Meier method.
Time Frame: Assessed from the date of study enrollment until death from any cause, or last follow-up, whichever occurs first, assessed up to 5 years from study enrollment
Reporting Status: Not Posted, anticipated posting 2026-01

11. Secondary Outcome: Phase 1: Event-free Survival (EFS)
Description: EFS is defined as the time from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), death, or last follow-up, whichever occurs first, assessed using the Kaplan-Meier method. Disease progression is an increase by ≥ 50% from progressive disease progression (PPD) nadir and an increase in longest transverse diameter of a lesion (LDi) or shortest axis perpendicular diameter (SDi) from nadir of >0.5 cm for lesions <2 cm or >1.0 cm for lesions >2 cm as assessed by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL).
Time Frame: Assessed from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), death, or last follow-up, whichever occurs first, assessed up to 8 months
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Months | 1.48 [0.49 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | 4.14 [2.99 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable. | 1.59 [0.66 to NA] — The confidence intervals (CI) are generated from the Brookmeyer-Crowley method, where if the estimate of a limit of a generated CI does not cross the median then it is reported as not estimable.

12. Other Pre Specified Outcome: Phase 1: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 24 cycles (i.e., 72 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
Number analyzed (Participants) | 3 | 3 | 2
Participants | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events was monitored/assessed 24 cycles (i.e., 72 weeks).
Arm/Group | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg (N=3) | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg (N=3) | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg (N=2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 1 Enitociclib (VIP152) 15 mg and Venetoclax 600 mg (N=3) | Cohort 1/Phase 1: Arm 1 Dose Escalation Dose Level 2 Enitociclib(VIP152) 22.5 mg & Venetoclax 600 mg (N=3) | Cohort 1/Phase 1:Arm 1 Dose Escalation Dose Level 3 Enitociclib (VIP152) 30 mg and Venetoclax 600 mg (N=2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (4) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (15) | 2 (13) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 2 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 3 (5) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 3 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 3 (13) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (7) | 2 (12) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Tinea corporis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT05371054/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT05371054/ICF_001.pdf